CLINICAL TRIAL: NCT00717405
Title: An Open Label Study to Assess the Rate of Pathological Complete Response in Patients With Primary Inflammatory HER2-positive Breast Cancer Treated With Avastin + Herceptin Based Chemotherapy
Brief Title: A Study of Avastin (Bevacizumab) Plus Herceptin (Trastuzumab) in Patients With Primary Inflammatory HER2-Positive Breast Cancer.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML21531; 2008-000783-16
Record Dates: First submitted 2008-07-16; First posted 2008-07-17 (Estimated); Results first posted 2016-01-06 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab; Trastuzumab

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Standard chemotherapy; Drug: bevacizumab [Avastin]; Drug: trastuzumab [Herceptin]

INTERVENTIONS:
Drug: Standard chemotherapy — As prescribed
Drug: bevacizumab [Avastin] — 15mg/kg iv 3 weekly in cycles 1-8
Drug: trastuzumab [Herceptin] — 8mg/kg iv loading dose followed by 6mg/kg iv 3 weekly in cycles 5-8.

SUMMARY:
This single arm study will assess the efficacy and safety of preoperative treatment with Avastin combined with Herceptin-based chemotherapy in patients with primary inflammatory HER2-positive breast cancer. Patients will be treated with a total of 8 cycles of pre-operative chemotherapy + Avastin + Herceptin. The anticipated time on study treatment is 3-12 months, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult females, >=18 years of age;
* inflammatory breast cancer;
* HER2-positive tumors;
* performance status 0-2.

Exclusion Criteria:

* metastases;
* previous treatment with chemotherapy, radiation therapy or hormone therapy for a breast tumor;
* clinically significant cardiovascular disease, or history of thrombotic disorders.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2008-10; Primary Completion 2010-04 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (25):
- France (25):
  - Besançon
  - Bordeaux
  - Brest
  - Caen
  - Clermont-Ferrand
  - Dijon
  - La Tronche
  - Lille
  - Lyon
  - Marseille
  - Montpellier
  - Nantes
  - Nice
  - Paris
  - Reims
  - Rennes
  - Rouen
  - Saint-Brieuc
  - Saint-Cloud
  - Saint-Herblain
  - Saint-Priest-en-Jarez
  - Strasbourg
  - Toulouse
  - Vandœuvre-lès-Nancy
  - Villejuif

REFERENCES:
- [Derived] Pierga JY, Petit T, Delozier T, Ferrero JM, Campone M, Gligorov J, Lerebours F, Roche H, Bachelot T, Charafe-Jauffret E, Pavlyuk M, Kraemer S, Bidard FC, Viens P. Neoadjuvant bevacizumab, trastuzumab, and chemotherapy for primary inflammatory HER2-positive breast cancer (BEVERLY-2): an open-label, single-arm phase 2 study. Lancet Oncol. 2012 Apr;13(4):375-84. doi: 10.1016/S1470-2045(12)70049-9. Epub 2012 Feb 28. PMID 22377126

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab + Trastuzumab Chemotherapy: Neoadjuvant treatment (Cycles 1-8, 3-week cycle): Participants received 15 milligrams per kilogram (mg/kg) intravenous (IV) bevacizumab every 3 weeks (q3w) for 8 cycles, 4 cycles of 500 milligrams per squared-meter (mg/m^2) IV 5-fluorouracil, 100 mg/m^2 IV epirubicin, and 500 mg/m^2 IV cyclophosphamide, q3w, followed by 4 cycles of 100 mg/m^2 IV docetaxel q3w plus trastuzumab (loading dose of 8 mg/kg and then 6 mg/kg q3w). Participants underwent surgery (mastectomy) after neoadjuvant treatment, maintaining trastuzumab (6 mg/kg). Adjuvant treatment: Participants received radiotherapy 2-4 weeks after surgery and lasted for 4-6 weeks, 6 mg/kg IV trastuzumab q3w and 15 mg/kg IV bevacizumab q3w administered along with/after the radiotherapy (administered up to a cumulative [neoadjuvant + adjuvant] total of 18 injections each. Hormonal therapy (at investigator discretion) after the end of radiotherapy was administered for 5 years, if participant was hormone receptor positive.
Period: Overall Study
Arm/Group | Bevacizumab + Trastuzumab Chemotherapy
Started | 52
Completed | 52
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Intent to treat population (ITT): Included all enrolled participants who had at least 1 post baseline assessment.
Groups:
- Bevacizumab + Trastuzumab: Neoadjuvant treatment (Cycles 1-8, 3-week cycle): Participants received 15 mg/kg IV bevacizumab q3w for 8 cycles, 4 cycles of 500 mg/m^2 IV 5-fluorouracil, 100 mg/m^2 IV epirubicin, and 500 mg/m^2 IV cyclophosphamide, q3w, followed by 4 cycles of 100 mg/m^2 IV docetaxel q3w plus trastuzumab (loading dose of 8 mg/kg and then 6 mg/kg q3w). Participants underwent surgery (mastectomy) after neoadjuvant treatment, maintaining trastuzumab (6 mg/kg). Adjuvant treatment: Participants received radiotherapy 2-4 weeks after surgery and lasted for 4-6 weeks, 6 mg/kg IV trastuzumab q3w and 15 mg/kg IV bevacizumab q3w administered along with/after the radiotherapy (administered up to a cumulative [neoadjuvant + adjuvant] total of 18 injections each. Hormonal therapy (at investigator discretion) after the end of radiotherapy was administered for 5 years, if participant was hormone receptor positive.
Arm/Group | Bevacizumab + Trastuzumab
Number analyzed (Participants) | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.48 (9.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Pathological Complete Response (PCR) According to the Sataloff Classification
Description: PCR was assessed at the time of definitive surgery according to Sataloff classification and centrally reviewed by an independent committee under blinded conditions. Pathological response was defined based on the therapeutic response at the primary tumor site and axillary lymph nodes. Primary tumor response criteria were as follows: T-A (Total / near total therapeutic effect), T-B (Subjectively greater than [>] 50 percent [%] therapeutic effect but less than [<] T-A), T-C (<50% therapeutic effect, but effect evident), T-D (No therapeutic effect). Axillary lymph node response: N-A (Evidence of therapeutic effect, no metastases), N-B (No therapeutic effect, no nodal metastases), N-C (Nodal metastasis but evident therapeutic effect), N-D (Nodal metastasis with no therapeutic effect). T-A and N-A or T-A and N-B responses were defined as PCR and all other tumor responses as non-responders. Participants with missing values were considered as non-responders.
Time Frame: From baseline through Week 25 (Up to 6 months)
Population: ITT population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab + Trastuzumab
Number analyzed (Participants) | 52
percentage of participants | 63.46 [49.41 to 77.51]

2. Secondary Outcome: Percentage of Participants With a PCR According to the Chevallier Classification
Description: PCR was assessed at the time of definitive surgery according to Chevallier classification and centrally reviewed by an independent committee under blinded conditions. The Chevallier classification for grading of therapeutic effect related to the primary tumor site and axillary lymph nodes was defined by microscopic changes as follows - Grade 1: Disappearance of all tumors either in the breast or in the nodes, Grade 2: Persistence of carcinoma in situ in the breast only and no nodal invasion, Grade 3: Presence of invasive carcinoma with stromal alteration, Grade 4: Presence of invasive carcinoma without modification. Grade 1 response was considered as PCR. Participants with missing values were considered as non-responders.
Time Frame: From baseline through Week 25 (Up to 6 months)
Population: ITT population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab + Trastuzumab
Number analyzed (Participants) | 52
percentage of participants | 53.85 [39.34 to 68.36]

3. Secondary Outcome: Percentage of Participants Who Were Responders Based on Inflammatory Signs From Baseline at Cycle 5 and Final Treatment Visit
Description: Breast tumor was physically evaluated during the study which included assessment for inflammatory signs and for overall clinical response. Participant with response from baseline based on inflammatory signs at Cycle 5 and final treatment visit were presented.
Time Frame: Baseline, Cycle 5 (Week 15), Neo-adjuvant treatment final visit (Week 25)
Population: ITT population. Number of participants analyzed included participants for whom tumor physical examination was performed and were evaluated for response from baseline assessment of inflammatory signs. n included number of participants who were evaluable at a particular time point.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + Trastuzumab
Number analyzed (Participants) | 43
percentage of participants
  Response from baseline at Week 15 (n=43) | 88.4
  Response from baseline at Week 25 (n=42) | 100.0

4. Secondary Outcome: Percentage of Participants Who Were Responders Based on Overall Clinical Response From Baseline at Cycle 5 and Final Treatment Visit
Description: Breast tumor was physically evaluated during the study which included assessment for inflammatory signs and for overall clinical response. Participant with response from baseline based on overall clinical response at Cycle 5 and final treatment visit were presented.
Time Frame: Baseline, Cycle 5 (Week 15), Neo-adjuvant treatment final visit (Week 25)
Population: ITT population. Number of participants analyzed included participants for whom tumor physical examination was performed. n included number of participants who were evaluable at a particular time point.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + Trastuzumab
Number analyzed (Participants) | 45
percentage of participants
  Response from baseline at Week 15 (n=44) | 90.9
  Response from baseline at Week 25 (n=45) | 97.8

5. Secondary Outcome: Number of Participants Who Underwent Mastectomy
Description: Surgery included a mastectomy with axillary node dissection and had to be performed at least 4 weeks after the last infusion of neoadjuvant bevacizumab treatment.
Time Frame: Anytime between Week 26 and Week 29
Population: ITT population.
Measure: Number; unit: participants
Arm/Group | Bevacizumab + Trastuzumab
Number analyzed (Participants) | 52
participants | 49

6. Secondary Outcome: Percentage of Participants With Macroscopically Visible Tumor
Description: Local pathologists assessed the tumor whether it was macroscopically visible or not and percentage of participants for whom the tumor was macroscopically visible was reported.
Time Frame: Anytime between Week 26 and Week 29
Population: ITT population. Included participants who underwent mastectomy.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + Trastuzumab
Number analyzed (Participants) | 49
percentage of participants | 26.5

7. Secondary Outcome: Percentage of Participants Who Underwent Lymph Node Resection
Description: Among the participants who were planned to undergo mastectomy, lymph node resection was also performed by the physician depending up on the participant's breast cancer grades.
Time Frame: Anytime between Week 26 and Week 29
Population: ITT population. Included participants who underwent mastectomy.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + Trastuzumab
Number analyzed (Participants) | 49
percentage of participants | 98.0

8. Secondary Outcome: Breast Cancer Marker CA15.3 at Baseline, Neoadjuvant Final Visit and Change From Baseline at Neoadjuvant Final Visit
Time Frame: Baseline, Neoadjuvant Final Visit (Week 25)
Population: Safety population: Number of participants included all the participants who received at least one infusion of bevacizumab. n included participants who were evaluable at that time point.
Measure: Mean (Standard Deviation); unit: Units per milliliter (U/mL)
Arm/Group | Bevacizumab + Trastuzumab
Number analyzed (Participants) | 52
Units per milliliter (U/mL)
  Baseline (n=52) | 39.66 (79.49)
  Neoadjuvant final visit (n=37) | 29.39 (10.06)
  Change in CA15.3 at neoadjuvant final visit (n=37) | -3.39 (33.05)

9. Secondary Outcome: Percentage of Participants Who Were Disease Free at 3 and 5 Years
Description: A participant was considered disease free if the participant did not experience any of the following events: local recurrence in the ipsilateral breast following lumpectomy, regional recurrence, distant recurrence, contralateral breast cancer, second primary cancer (other than squamous or basal cell carcinoma of the skin, melanoma in situ, carcinoma in situ of the cervix, colon carcinoma in situ, or lobular carcinoma in situ of the breast), or death from any cause.
Time Frame: 3, 5 years
Population: ITT population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab + Trastuzumab
Number analyzed (Participants) | 52
percentage of participants
  3 years | 66.7 [52.0 to 77.8]
  5 years | 60.8 [46.1 to 72.7]

10. Secondary Outcome: Disease Free Survival (DFS) Duration
Description: DFS was estimated using Kaplan-Meier method.
Time Frame: Up to 5 Years
Population: ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab + Trastuzumab
Number analyzed (Participants) | 52
months | NA [NA to NA] — Using Kaplan-Meier method, median DFS was not reached due to higher (>50%) number of censored participants.

11. Secondary Outcome: Percentage of Participants Who Were Recurrence Free at 3 and 5 Years
Description: A participant was considered recurrence free if the participant did not experience local or regional recurrence (wall or axillaries nodes), or occurrence of distant metastases (including soft tissue and distal lymph nodes).
Time Frame: 3, 5 years
Population: ITT population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab + Trastuzumab
Number analyzed (Participants) | 52
percentage of participants
  3 years | 69.7 [54.8 to 80.5]
  5 years | 65.4 [50.4 to 76.9]

12. Secondary Outcome: Recurrence Free Survival (RFS) Duration
Description: RFS was estimated using Kaplan-Meier method.
Time Frame: Up to 5 Years
Population: ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab + Trastuzumab
Number analyzed (Participants) | 52
months | NA [NA to NA] — Using Kaplan-Meier method, median RFS was not reached due to higher (>50%) number of censored participants.

13. Secondary Outcome: Percentage of Participants Who Were Alive at 3 and 5 Years
Time Frame: 3, 5 years
Population: ITT population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab + Trastuzumab
Number analyzed (Participants) | 52
percentage of participants
  Alive at 3 years | 90.0 [77.6 to 95.7]
  Alive at 5 years | 81.8 [67.9 to 90.1]

14. Secondary Outcome: Overall Survival (OS) Duration
Description: OS was defined as the time from the first administration of neoadjuvant treatment to death of any cause. OS was estimated using Kaplan-Meier method.
Time Frame: Up to 5 years
Population: ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab + Trastuzumab
Number analyzed (Participants) | 52
months | NA [NA to NA] — Using Kaplan-Meier method, Median OS was not reached due to higher (>50%) number of censored participants

ADVERSE EVENTS:
Time Frame: From Baseline until end of study (Up to approximately 6 years)
Arm/Group | Bevacizumab + Trastuzumab
Serious Adverse Events (participants affected / at risk) | 20/52
Other Adverse Events (participants affected / at risk) | 52/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + Trastuzumab (N=52)
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 5
Febrile neutropenia (Blood and lymphatic system disorders) | 6
Vomiting (Gastrointestinal disorders) | 1
Hyperthermia (General disorders) | 1
Malaise (General disorders) | 1
Pyrexia (General disorders) | 1
Anal abscess (Infections and infestations) | 2
Appendicitis (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Ejection fraction decreased (Investigations) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Metrorrhagia (Reproductive system and breast disorders) | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Jugular vein thrombosis (Vascular disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 6
Atrial tachycardia (Cardiac disorders) | 1
Tooth loss (Gastrointestinal disorders) | 1
Impaired healing (General disorders) | 3
Inflammation (General disorders) | 1
Incision site abscess (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1
Nasal septum perforation (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 1
Lymphocele (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + Trastuzumab (N=52)
Anaemia (Blood and lymphatic system disorders) | 8
Febrile neutropenia (Blood and lymphatic system disorders) | 11
Leukopenia (Blood and lymphatic system disorders) | 7
Neutropenia (Blood and lymphatic system disorders) | 24
Cardiac failure congestive (Cardiac disorders) | 10
Conjunctivitis (Eye disorders) | 12
Lacrimation increased (Eye disorders) | 13
Abdominal pain (Gastrointestinal disorders) | 3
Abdominal pain upper (Gastrointestinal disorders) | 11
Constipation (Gastrointestinal disorders) | 14
Diarrhoea (Gastrointestinal disorders) | 9
Dyspepsia (Gastrointestinal disorders) | 6
Dysphagia (Gastrointestinal disorders) | 6
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 8
Gingival bleeding (Gastrointestinal disorders) | 8
Gingivitis (Gastrointestinal disorders) | 5
Haemorrhoids (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 36
Vomiting (Gastrointestinal disorders) | 18
Asthenia (General disorders) | 41
Fatigue (General disorders) | 4
Mucosal inflammation (General disorders) | 34
Oedema peripheral (General disorders) | 6
Pyrexia (General disorders) | 10
Bronchitis (Infections and infestations) | 8
Nasopharyngitis (Infections and infestations) | 8
Oral fungal infection (Infections and infestations) | 4
Pharyngitis (Infections and infestations) | 5
Rhinitis (Infections and infestations) | 9
Tonsillitis (Infections and infestations) | 6
Tooth abscess (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 6
Radiation skin injury (Injury, poisoning and procedural complications) | 19
Gamma-glutamyltransferase increased (Investigations) | 5
Weight decreased (Investigations) | 6
Anorexia (Metabolism and nutrition disorders) | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 15
Back pain (Musculoskeletal and connective tissue disorders) | 8
Bone pain (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 13
Ageusia (Nervous system disorders) | 5
Dysgeusia (Nervous system disorders) | 8
Headache (Nervous system disorders) | 17
Neuropathy peripheral (Nervous system disorders) | 10
Anxiety (Psychiatric disorders) | 4
Insomnia (Psychiatric disorders) | 4
Proteinuria (Renal and urinary disorders) | 32
Breast pain (Reproductive system and breast disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 33
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 7
Alopecia (Skin and subcutaneous tissue disorders) | 36
Dry skin (Skin and subcutaneous tissue disorders) | 9
Erythema (Skin and subcutaneous tissue disorders) | 16
Nail toxicity (Skin and subcutaneous tissue disorders) | 7
Onycholysis (Skin and subcutaneous tissue disorders) | 10
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 9
Skin exfoliation (Skin and subcutaneous tissue disorders) | 5
Skin toxicity (Skin and subcutaneous tissue disorders) | 4
Hypertension (Vascular disorders) | 21
Vertigo (Ear and labyrinth disorders) | 6
Oesophagitis (Gastrointestinal disorders) | 4
Chest pain (General disorders) | 4
Pain (General disorders) | 3
Hot flush (Vascular disorders) | 7
Lymphocele (Vascular disorders) | 15
Lymphoedema (Vascular disorders) | 10
Cystitis (Infections and infestations) | 4
Sinusitis (Infections and infestations) | 4
Skin infection (Infections and infestations) | 5
Tooth infection (Infections and infestations) | 4
Wound dehiscence (Injury, poisoning and procedural complications) | 4
Ejection fraction decreased (Investigations) | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 5
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Neuralgia (Nervous system disorders) | 4
Paraesthesia (Nervous system disorders) | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Dermatitis (Skin and subcutaneous tissue disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 4
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 4
Rectal hemorrhage (Gastrointestinal disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.